CLINICAL TRIAL: NCT03773575
Title: Evaluation of Closed Incision Negative Pressure Dressing (PREVENA) to Prevent Lower Extremity Amputation Wound Complications
Acronym: PREVENA-AMP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Acelity (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 18P.577
Record Dates: First submitted 2018-12-10; First posted 2018-12-12 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Amputation; Amputation; Postoperative, Sequelae; Wound Dehiscence; Seroma; Wound Infection, Surgical; Lymph Leakage
MeSH Terms: conditions — Seroma; Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Prevena (Experimental): PREVENA™ PEEL & PLACE™ Dressing Kit
  Interventions: Device: PREVENA™ PEEL & PLACE™ Dressing Kit
- Standard Care (No Intervention): sterile gauze dressing supplemented with an Ace wrap

INTERVENTIONS:
Device: PREVENA™ PEEL & PLACE™ Dressing Kit — In combination with a negative pressure pump (V.A.C. ® Therapy Unit, KCI USA, Inc.), the Prevena dressing is designed to provide negative pressure wound therapy (NPWT) over surgical incisions (incisional NPWT).
  Arms: Prevena

SUMMARY:
This study is a prospective, multi-center, two-arm, unblinded, and randomized controlled trial with a goal of evaluating the impact of a closed incision negative pressure dressing (PREVENA) on incidence of post-operative wound complications and medical costs in patients undergoing lower extremity amputation.

DETAILED DESCRIPTION:
This is a prospective, multi-center, two-arm, unblinded, randomized controlled trial to evaluate the impact of a closed incision negative pressure dressing (PREVENA™ PEEL & PLACE™ Dressing Kit) on incidence of post-operative wound complications in patients undergoing above-the-knee (AKA) or below-the-knee (BKA) amputation. Up to 440 subjects at approximately five (5) participating sites will be randomized to receive either the Prevena dressing or a standard care dressing. The incision will be assessed for complications at post-op day 5 or day 6 and at approximately 30 days after discharge. The primary outcome of this study is reported wound complications, including dehiscence (opening of the incision), seroma, lymph leak, infection (deep or superficial), hematoma (blood clots), ischemia (decreased blood supply), and necrosis (tissue death) A major complication is defined as any wound complication requiring intravenous or oral antibiotics, reoperation and/or hospital readmission. All data (demographics, medical history, and clinical outcomes) will be collected via medical record review

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults 18 years or older
2. Patients undergoing above-knee amputation (includes the revision of emergency guillotine amputations)
3. Patients undergoing below-knee amputation (includes the revision of emergency guillotine amputations)
4. Informed Consent signed by patient

Exclusion Criteria:

1. Minors under 18 years
2. Women who are pregnant or breastfeeding
3. Patients undergoing emergent or guillotine amputation
4. Patients having BOTH legs amputated
5. Patients with sensitivity to silver
6. Unwilling or unable to provide informed consent
7. Inability to comply with planned study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 272 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-08-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul DiMuzio, MD, Principal Investigator — Thomas Jefferson University
Locations (3):
- United States (2):
  - Westchester Medical Center, Valhalla, New York
  - Thomas Jefferson University/Hospital, Philadelphia, Pennsylvania
- Gemelli Hospital, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasanadka R, McLafferty RB, Moore CJ, Hood DB, Ramsey DE, Hodgson KJ. Predictors of wound complications following major amputation for critical limb ischemia. J Vasc Surg. 2011 Nov;54(5):1374-82. doi: 10.1016/j.jvs.2011.04.048. Epub 2011 Aug 15. PMID 21840153
- [Background] Belmont PJ Jr, Davey S, Orr JD, Ochoa LM, Bader JO, Schoenfeld AJ. Risk factors for 30-day postoperative complications and mortality after below-knee amputation: a study of 2,911 patients from the national surgical quality improvement program. J Am Coll Surg. 2011 Sep;213(3):370-8. doi: 10.1016/j.jamcollsurg.2011.05.019. Epub 2011 Jul 1. PMID 21723151
- [Background] Stannard JP, Volgas DA, McGwin G 3rd, Stewart RL, Obremskey W, Moore T, Anglen JO. Incisional negative pressure wound therapy after high-risk lower extremity fractures. J Orthop Trauma. 2012 Jan;26(1):37-42. doi: 10.1097/BOT.0b013e318216b1e5. PMID 21804414
- [Background] Pachowsky M, Gusinde J, Klein A, Lehrl S, Schulz-Drost S, Schlechtweg P, Pauser J, Gelse K, Brem MH. Negative pressure wound therapy to prevent seromas and treat surgical incisions after total hip arthroplasty. Int Orthop. 2012 Apr;36(4):719-22. doi: 10.1007/s00264-011-1321-8. Epub 2011 Jul 15. PMID 21761149
- [Background] Grauhan O, Navasardyan A, Hofmann M, Muller P, Stein J, Hetzer R. Prevention of poststernotomy wound infections in obese patients by negative pressure wound therapy. J Thorac Cardiovasc Surg. 2013 May;145(5):1387-92. doi: 10.1016/j.jtcvs.2012.09.040. Epub 2012 Oct 27. PMID 23111014
- [Background] Hyldig N, Birke-Sorensen H, Kruse M, Vinter C, Joergensen JS, Sorensen JA, Mogensen O, Lamont RF, Bille C. Meta-analysis of negative-pressure wound therapy for closed surgical incisions. Br J Surg. 2016 Apr;103(5):477-86. doi: 10.1002/bjs.10084. PMID 26994715
- [Background] Kwon J, Staley C, McCullough M, Goss S, Arosemena M, Abai B, Salvatore D, Reiter D, DiMuzio P. A randomized clinical trial evaluating negative pressure therapy to decrease vascular groin incision complications. J Vasc Surg. 2018 Dec;68(6):1744-1752. doi: 10.1016/j.jvs.2018.05.224. Epub 2018 Aug 17. PMID 30126781
- [Background] O'Brien PC, Fleming TR. A multiple testing procedure for clinical trials. Biometrics. 1979 Sep;35(3):549-56. PMID 497341
- See also: National Healthcare Safety Network definition of Surgical Site Infection (SSI) Event — http://www.cdc.gov/nhsn/PDFs/pscManual/9pscSSIcurrent.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prevena | Standard Care
Started | 137 | 135
Completed | 134 | 129
Not Completed | 3 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prevena | Standard Care | Total
Number analyzed (Participants) | 134 | 129 | 263
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (13) | 64 (11) | 65 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 42 | 82
  Male | 94 | 87 | 181
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 42 | 37 | 79
  White | 86 | 85 | 171
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 13 | 21
  Not Hispanic or Latino | 117 | 103 | 220
  Unknown or Not Reported | 9 | 13 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Wound Complications
Description: Presence of any of the following post-procedure:
  * Dehiscence (skin or fascia)
  * Seroma
  * Lymph leak
  * Infection (superficial or deep, using CDC Surgical Site Infection criteria)
  * Hematoma
  * Ischemia
  * Necrosis
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 26 | 31

2. Secondary Outcome: Length of Stay (LOS)
Description: index LOS is defined as days from operation to discharge; 30d LOS is defined as the index LOS plus all readmission days within 30d related to any wound complication
Time Frame: 30 days post procedure
Measure: Mean (Standard Deviation); unit: Length of stay in days
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Length of stay in days | 10 (7.6) | 9.6 (6.5)

3. Secondary Outcome: 30-day Return to Operating Room (ROR)
Description: Reoperation for wound complication within 30 days involving incision and drainage in the operating room; opening the skin to drain a superficial soft tissue infection at bedside or in the office is not considered reoperation
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 5 | 11

4. Secondary Outcome: 30-day Hospital Readmissions
Description: Rehospitalization for wound complication within 30 days
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 12 | 15

5. Secondary Outcome: Incidence of Skin Dehiscence
Description: Individual rates of the incidence of skin dehiscence
Time Frame: 30 days post procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 15 | 11

6. Secondary Outcome: Incidence of Fascial Dehiscence
Description: Individual incidence rate of fascial dehiscence
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 2 | 2

7. Secondary Outcome: Incidence of Superficial Skin Infection
Description: Individual incidence of superficial skin infection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 2 | 2

8. Secondary Outcome: Incidence of Deep Skin Infection
Description: Individual incidence of deep skin infection
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 5 | 4

9. Secondary Outcome: Incidence of Seroma
Description: Individual incidence of seroma
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 1 | 1

10. Secondary Outcome: Incidence of Hematoma
Description: Individual Incidence of Hematoma
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 2 | 3

11. Secondary Outcome: Incidence of Necrosis
Description: Individual incidence of Necrosis
Time Frame: 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Prevena | Standard Care
Number analyzed (Participants) | 134 | 129
Participants | 4 | 10

ADVERSE EVENTS:
Time Frame: 30 days following hospitalization for amputation
Arm/Group | Prevena | Standard Care
All-Cause Mortality (participants affected / at risk) | 1/134 | 1/129
Serious Adverse Events (participants affected / at risk) | 11/134 | 14/129
Other Adverse Events (participants affected / at risk) | 0/134 | 0/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prevena (N=134) | Standard Care (N=129)
Sepsis (Immune system disorders) | 2 (2) | 0 (0)
Skin Dehiscence (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Delayed Wound Healing (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Hematoma (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Homorrhage from Operative Site (Vascular disorders) | 0 (0) | 2 (2)
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Loose Staple (Product Issues) | 1 (1) | 0 (0) — Loose staple after trauma to surgical site
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Worsening post-procedure pain (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Angina (Cardiac disorders) | 1 (1) | 0 (0)
Acute respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Soft Tissue Infection (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
STEMI (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/75/NCT03773575/Prot_SAP_000.pdf